CLINICAL TRIAL: NCT04968353
Title: Effect of Clear Aligner Attachment Design on Extrusion of Maxillary Lateral Incisors: a Randomized Prospective Clinical Trial
Brief Title: Effect of Clear Aligner Attachment Design on Extrusion of Maxillary Lateral Incisors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HM20021396
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Maxillary Lateral Incisor Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Incisally-beveled (Active Comparator): Use of incisally-beveled attachment to extrude lateral incisor
  Interventions: Device: Incisally-beveled attachment
- Gingivally-beveled (Active Comparator): Use of gingivally-beveled attachment to extrude lateral incisor
  Interventions: Device: Gingivally-beveled attachment
- Optimized (Active Comparator): Use of optimized attachment to extrude lateral incisor
  Interventions: Device: Optimized attachment
- Horizontal (Active Comparator): Use of horizontal (unbeveled) attachment to extrude lateral incisor
  Interventions: Device: Horizontal attachment

INTERVENTIONS:
Device: Incisally-beveled attachment — Incisally-beveled attachments will be bonded to teeth before or during orthodontal treatment with clear aligners
  Arms: Incisally-beveled
Device: Gingivally-beveled attachment — Gingivally-beveled attachments will be bonded to teeth before or during orthodontal treatment with clear aligners
  Arms: Gingivally-beveled
Device: Optimized attachment — Optimized attachments will be bonded to teeth before or during orthodontal treatment with clear aligners
  Arms: Optimized
Device: Horizontal attachment — Horizontal attachments will be bonded to teeth before or during orthodontal treatment with clear aligners
  Arms: Horizontal

SUMMARY:
The purpose of this research is to test which of four clear aligner attachment types is more efficient in extruding (erupting) maxillary lateral incisors vertically into correct position during orthodontic treatment.

DETAILED DESCRIPTION:
Attachments are small tooth-colored shapes that are bonded (attached) to teeth before or during treatment with clear aligners. They are like handles, giving aligners something to gently push teeth into correct positions. There are 4 different shapes of attachments that are commonly used to extrude lateral incisors (incisally-beveled, gingivally-beveled, optimized and horizontal). All 4 of these attachments are successful in extruding lateral incisors but there is not enough research evidence to know for sure which attachment would be ideal for a specific circumstance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 16 years or older to be treated with either Comprehensive Invisalign or Invisalign Teen,
2. Maxillary lateral incisor requiring 0.3 mm or more extrusion (as determined by ClinCheck),
3. Maxillary arch with less than 6 mm of crowding or spacing,
4. All teeth present and fully erupted (excluding third molars).

Exclusion Criteria:

1. Presence of anterior crossbite
2. Any missing teeth in the maxillary arch
3. Treatment plan includes surgery or extraction of any maxillary teeth,
4. Maxillary lateral incisors with pathology or large restorations (crowns)
5. Maxillary lateral incisors have a less than 0.3 mm of extrusion prescribed in the Tooth Movement Table on the Invisalign ClinCheck

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindauer, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Groody JT, Lindauer SJ, Kravitz ND, Carrico CK, Madurantakam P, Shroff B, Darkazanli M, Gardner WG. Effect of clear aligner attachment design on extrusion of maxillary lateral incisors: A multicenter, single-blind randomized clinical trial. Am J Orthod Dentofacial Orthop. 2023 Nov;164(5):618-627. doi: 10.1016/j.ajodo.2023.07.011. Epub 2023 Aug 21. PMID 37610383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began August, 2021 and final data collection was completed in June, 2022. Patients were recruited from 3 orthodontic practices. Units enrolled are counted as numbers of teeth. Potentially, 2 maxillary lateral incisors from each patient could have been enrolled.
Units Other Than Participants: Teeth
Period: Overall Study
Arm/Group | Horizontal | Incisally-beveled | Gingivally-beveled | Optimized
Started | 20; 20 Teeth | 15; 15 Teeth | 16; 16 Teeth | 22; 23 Teeth
Completed | 19; 19 Teeth | 15; 15 Teeth | 14; 14 Teeth | 22; 23 Teeth
Not Completed | 1; 1 Teeth | 0; 0 Teeth | 2; 2 Teeth | 0; 0 Teeth
Not completed — Non-compliance | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Incisally-beveled | Gingivally-beveled | Optimized | Horizontal | Total
Number analyzed (Participants) | 15 | 14 | 22 | 19 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 9 | 8 | 20
  Between 18 and 65 years | 12 | 12 | 13 | 11 | 48
  >=65 years | 1 | 1 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (15.3) | 31.2 (15.6) | 32.1 (14.26) | 30.4 (15.16) | 31.3 (15.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 14 | 13 | 49
  Male | 3 | 4 | 8 | 6 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 2 | 6
  Asian | 3 | 3 | 3 | 2 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 3 | 8
  White | 9 | 9 | 15 | 12 | 45
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 22 | 20 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percent of Vertical Tooth Movement
Description: Percent achieved of the vertical (inciso-gingival) tooth movement will be assessed by comparing the initial ClinCheck software estimate tooth movement required to the amount of tooth movement observed
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: percentage of predicted
Units Other Than Participants: Teeth
Arm/Group | Horizontal | Incisally-beveled | Gingivally-beveled | Optimized
Number analyzed (Participants) | 19 | 15 | 14 | 22
Number analyzed (Teeth) | 19 | 15 | 14 | 23
percentage of predicted | 79 [58 to 100] | 78 [58 to 98] | 78 [63 to 93] | 62 [40 to 84]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Horizontal | Incisally-beveled | Gingivally-beveled | Optimized
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/14 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/14 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/14 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04968353/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT04968353/ICF_001.pdf